CLINICAL TRIAL: NCT02811185
Title: An Open-label, Non-randomized Study to Monitor for Adverse Drug Reactions Among Patients Administered Fedoruk-manufactured [F-18]-FDG Injection
Brief Title: Registry Type Study to Monitor for Adverse Drug Reactions to Fedoruk Manufactured [F-18]-Fludeoxyglucose
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Sylvia Fedoruk Canadian Centre for Nuclear Innovation (Other); Saskatoon Health Region (Other)
Responsible Party: Principal Investigator, Paul Babyn, M.D., University of Saskatchewan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FED001
Record Dates: First submitted 2016-06-15; First posted 2016-06-23 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Positron-Emission Tomography and Cone-Beam Computed Tomography
Keywords: PET; CT; PET/CT
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PET/CT Scan (Other): Subjects will receive a single dose of [F-18]-FDG Injection at Visit 1, followed by PET/CT scanning according to departmental practice.
  Interventions: Drug: [F-18]-Fludeoxyglucose
- PET Scan (Other): Subjects will receive a single dose of [F-18]-FDG Injection at Visit 1, followed by PET scanning according to departmental practice.
  Interventions: Drug: [F-18]-Fludeoxyglucose

INTERVENTIONS:
Drug: [F-18]-Fludeoxyglucose — Radiopharmaceutical imaging agent
  Other Names: FDG; Fluorodeoxyglucose; F-18-FDG

SUMMARY:
This is a single-centre, open-label, non-randomized clinical trial designed to monitor the occurrence of adverse events associated with [F-18]-FDG Injection manufactured by the Fedoruk Centre. [F-18]-FDG Injection used in this clinical trial will be identical to commercial [F-18]-FDG that is already used at Royal University Hospital (RUH).

DETAILED DESCRIPTION:
This study will document the use of Fedoruk-manufactured [F-18]-FDG Injection (citrate formulation) in patients referred for [F-18]-FDG PET or PET/CT imaging at Royal University Hospital (RUH) in Saskatoon, SK. This investigational agent is produced using procedures, raw materials, equipment and quality standards that are equivalent to commercially-approved [F-18]-FDG Injection (Glucovision®, manufactured by the CPDC in Hamilton ON).

This is a single-centre, open-label, non-randomized study to monitor for adverse drug reactions among subjects administered Fedoruk-manufactured [F-18]-FDG Injection. Eligible subjects are those who would normally be referred by their physician for [F-18]-FDG PET or PET/CT imaging at RUH in Saskatoon, SK.

The primary goal of this study is to permit immediate access, with appropriate regulatory and REB oversight, to Fedoruk-manufactured [F-18]-FDG Injection pending commercial approval.

Monitoring for adverse drug reactions, during and after subjects are administered Fedoruk-manufactured [F-18]-FDG Injection, will support the primary objective of this study. Based on the well-established safety profile of [F-18]-FDG and the comparability of Fedoruk-manufactured [F-18]-FDG Injection to commercially-approved [F-18]-FDG Injection (Glucovision®), it is not expected that any ADRs will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Referred by treating physician to receive [F-18]-FDG and PET or PET/CT imaging;
* Meets all current local clinical criteria for receiving [F-18]-FDG and PET or PET/CT imaging;
* Ability to understand and the willingness to sign, or (in the case of paediatric patients) a parent/guardian who understands and is willing to sign, a written informed consent document;

Exclusion Criteria:

* Pregnant women; all women of child-bearing potential will have a confirmed negative urine pregnancy test prior to administration of [F-18]-FDG Injection;
* Subjects unwilling or unable to stop breast feeding for 24 hours;
* Subjects who are medically unstable, based on the Principal Investigator's assessment

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Document any adverse drug reactions, following administration of [F-18]-FDG Injection. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Rakheja, MD, Principal Investigator — Saskatoon Health Region